CLINICAL TRIAL: NCT05367986
Title: Lectro-acupuncture at Zusanli, Qihai, and Guanyuan Acupoints Regulate Immune Function in Patients With Sepsis
Brief Title: Electro-acupuncture at Zusanli, Qihai, and Guanyuan Acupoints Regulate Immune Function in Patients With Sepsis
Acronym: EAIm-sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Guang Yang, Director, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EAIm-sepsis
Record Dates: First submitted 2022-03-26; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; Immune Dysfunction
Keywords: Sepsis; Immune Dysfunction; Electro-acupuncture
MeSH Terms: conditions — Sepsis; Immune System Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western medicine group(WM group) (No Intervention): Patients in the Western medicine group received conventional treatment with Western medicine. According to International Guidelines for Management of Sepsis and Septic Shock: 2016, conventional treatment includes antibiotics and other anti-infection measures, fluid management, mechanical ventilation, and nutritional support, but does not include the use of immunosuppressants or immune enhancers including hormones, gamma globulin, and thymosin.
- electro-acupuncture (EA) group (Experimental): Patients in the electro-acupuncture group were treated with Western medicine and electro-acupuncture. Electro-acupuncture was given at the Zusanli (ST36), Guanyuan (CV4), and Qihai (CV6) acupoints, twice a day for 30 minutes, and for 5 days in total.
  Interventions: Device: electro-acupuncture

INTERVENTIONS:
Device: electro-acupuncture — Electro-acupuncture was given at the Zusanli (ST36), Guanyuan (CV4), and Qihai (CV6) acupoints, twice a day for 30 minutes, and for 5 days in total.
  1. Acupoints were selected as follows. (1) Zusanli (ST36) belongs to zuyangming stomach meridian. It is located on the anterolateral part of the lower leg 3 inches (4 horizontal fingers) below the eye of the external knee between the fibula and the tibia, and a horizontal finger (middle finger) width from the front edge of the tibia. (2) Guan yuan (CV4) is located 3 inches below the umbilicus, on the midline of the abdomen. (3) Qihai (CV6) is located 1.5 inches below the umbilicus on the midline.
  2. Acupuncture and electro-acupuncture methods were performed as follows. Participants were in the supine position, and needles was inserted in the skin . After the participant has acid, numbness, swelling, pain or other feelings, the electro-acupuncture device was connect to the acupuncture needle, the frequency was set to continuous wave.
  Arms: electro-acupuncture (EA) group

SUMMARY:
The purpose of this study was to investigate the biochemical and clinical effects of electro-acupuncture in patients with sepsis.

DETAILED DESCRIPTION:
Patients were randomly divided into an electro-acupuncture (EA) group and a Western medicine group(WM group) using restricted block randomization (1:1 ratio).

Patients in the Western medicine group received conventional treatment with Western medicine. According to the International Guidelines for Management of Sepsis and Septic Shock: 2016, conventional treatment includes antibiotics and other anti-infection measures, fluid management, mechanical ventilation, and nutritional support, but did not include the use of immunosuppressants or immune enhancers including hormones, gamma globulin, and thymosin. Patients in the electro-acupuncture group were treated with Western medicine and electro-acupuncture. Electro-acupuncture was given at the Zusanli (ST36), Guanyuan (CV4), and Qihai (CV6) acupoints, twice a day for 30 minutes, and for 5 days in total.

The indicators of immune dysfunction including the percentage of T lymphocyte subsets, percentage of natural killer (NK) cells, and serum soluble programed cell death protein (sPD-1) level, and clinical effect including APACHE-II and SOFA score, whole blood analysis, levels of tumor necrosis factor-α (TNF-α) and C-reactive protein (CRP), were determined before treatment and after treatment for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sepsis;
* Signed the informed consent form.

Exclusion Criteria:

* Pregnancy or psychiatric disorder;
* Immune deficiency or using immunosuppressants or immune enhancers;
* History of malignancy;
* HIV positive;
* Unwilling to participate in the study or cooperate with the treatment. Patients who cannot tolerate electroacupuncture treatment or loss of follow-up for complicating with other diseases during the study would be dropped off.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Proportion of T lymphocyte subsets(%) | 5 days after treatment was begun (at the 6th day)
  Detect proportion of CD3-T lymphocyte and CD4-T lymphocyte(%) in total T lymphocytes in blood by flow cytometry .
Proportion of natural killer(NK) cells(%) | 5 days after treatment was begun (at the 6th day)
  Detect proportion of NK cells in total lymphocytes in blood by flow cytometry.
Level of sPD-1 level(pg/ml) | 5 days after treatment was begun (at the 6th day)
  Serum soluble programed cell death protein (sPD-1) level in blood was measured with ELISA.

SECONDARY OUTCOMES:
Neutrophils/Lymphocytes(N/L) ratio(%) | 5 days after treatment was begun (at the 6th day)
  N/L ratio was defined as the ratio of neutrophils to lymphocytes. Whole blood analyzer was used to measure the count neutrophils and lymphocytes in the patient's blood, and calculate the ratio of neutrophil to lymphocyte count.
Level of C-reactive protein (CRP) (mg/L) | 5 days after treatment was begun (at the 6th day)
  Serum soluble CRP level in blood was measured with ELISA.
Level of Tumor necrosis factor-α (TNF-α) (pg/ml) | 5 days after treatment was begun (at the 6th day)
  Serum soluble TNF-α level in blood was measured with ELISA.
Acute Physiology and Chronic Health Evaluation-Ⅱ(APACHE-Ⅱ) score | 5 days after treatment was begun (at the 6th day)
  APACHE-Ⅱ score is used to evaluate the severity and prognosis of sepsis patients. Possible score range from 0 (the disease is mild and the prognosis is good) to 71(the disease is serious and the prognosis is poor).
Sequential Organ Failure Assessment (SOFA) score | 5 days after treatment was begun (at the 6th day)
  SOFA score is used to evaluate the severity of organ failure. Possible score range from 0 (organ failure is rare and mild) to 48(multiple organ failure, and it's serious).

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yang, Study Director — The Second Affiliated Hospital of Guangzhou University of Chinese Medicine
Locations (1):
- 2nd Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available on request from the corrresponding author.The data are not publicly available due to privacy or ethical restrictions.The data that supprot the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 1, 2023
Access Criteria: 1. Doctor or medical researcher
  2. Sign relevant confidentiality agreement.

REFERENCES:
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Hotchkiss RS, Monneret G, Payen D. Sepsis-induced immunosuppression: from cellular dysfunctions to immunotherapy. Nat Rev Immunol. 2013 Dec;13(12):862-74. doi: 10.1038/nri3552. Epub 2013 Nov 15. PMID 24232462
- [Background] Bosmann M, Ward PA. The inflammatory response in sepsis. Trends Immunol. 2013 Mar;34(3):129-36. doi: 10.1016/j.it.2012.09.004. Epub 2012 Oct 2. PMID 23036432
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Yang G, Hu RY, Deng AJ, Huang Y, Li J. Effects of Electro-Acupuncture at Zusanli, Guanyuan for Sepsis Patients and Its Mechanism through Immune Regulation. Chin J Integr Med. 2016 Mar;22(3):219-24. doi: 10.1007/s11655-016-2462-9. Epub 2016 Jan 29. PMID 26825083